CLINICAL TRIAL: NCT02057315
Title: A Randomized, Double-Blind, Cross-Over, Placebo-Controlled Study to Determine the Efficacy and Safety of ELS-M11 in Acute Migraine
Brief Title: Study to Determine the Efficacy and Safety of ELS-M11 in Acute Migraine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Achelios Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACH10200
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Migraine Headaches
Keywords: Migraine headache; Photophobia; Phonophobia; Aura; Topical treatment
MeSH Terms: conditions — Migraine Disorders; Photophobia; Hyperacusis; Epilepsy | interventions — Ketoprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ELS-M11 (Experimental): Topical 5% ELS-M11 (3 g)
  Interventions: Drug: ELS-M11; Drug: Placebo
- Placebo (Placebo Comparator): A matching formulation with no active ingredient
  Interventions: Drug: ELS-M11; Drug: Placebo

INTERVENTIONS:
Drug: ELS-M11 — One dose of 5% ELS-M11 over 3 bilateral applications.
  Other Names: Topofen (ketoprofen) Gel 5%
Drug: Placebo — One dose of matching placebo over 3 bilateral applications.

SUMMARY:
This is a Phase 1/ Phase 2, 12-week, multi-center, randomized, double-blind, cross-over, placebo-controlled study to evaluate the efficacy and safety of ELS-M11 compared to placebo in 50 male and female subjects, aged 18 to 65 years that suffer recurring moderate-severe migraine headaches (2-8 per month).

This study is designed to describe the efficacy and safety of ELS-M11 as compared to placebo.

DETAILED DESCRIPTION:
Achelios is developing ELS-M11 for topical application for the acute treatment of migraine events in patients with a history of migraine with or without aura.

To be eligible for the study, patients must have a one-year documented history of migraine headache (as defined by the International Headache Society IHS), with or without aura, with 2≤8 moderate or severe migraine attacks per month in the 2 months prior to the screening visit.

The total duration of the study is the completion of five migraine headaches per subject over a maximum 12 week period followed by a 3-14 day Follow-Up Period.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Males and females aged 18-65 who can read, write and understand English
* Subject has at least a one year documented history of migraine headache (defined by International headache Society IHS) migraine definitions, with or without aura, with 2≤8 moderate or severe migraine attacks per month in the 2 months prior to the screening visit
* Is stable on the current standard non-opioid rescue medication for at least 2 months prior to randomization
* Can distinguish migraine from tension headache (HA), with 24 hours of freedom from HA between migraine events
* Women of childbearing potential must be currently using or willing to use contraception (30 days prior to start of study medication and for 21 days after taking study medication)
* Women of non-childbearing potential include females regardless of age, with functioning ovaries and who have a current documented tubal ligation [Hatcher, 2004] bilateral oophorectomy or total hysterectomy, or post-menopausal females
* The subject is able and willing to perform the assessments and procedures as specified in this protocol, including the ability to learn and follow instructions for ePRO device

Exclusion Criteria:

* Migraineurs taking opioid-based rescue medications for any indication
* Subject has history of mild migraine events or migraines that usually resolve spontaneously in less than 2 hours
* Subject has menstrual migraines
* Positive Drug Test
* Subject has basilar or hemiplegic migraines
* Subject has more than 15 headache-days per month
* Subjects with a history of facial allodynia
* Subject has a history of vomiting during more than 30% of migraine episodes
* Self confinement to bed rest for more than 50% of migraine episodes
* Subject was greater than 50 years old at age of migraine onset
* Acute coronary syndrome (i.e., myocardial infarction and unstable angina), stroke or resuscitated cardiac arrest within the past 3 months
* Severe congestive heart failure
* Systolic blood pressure (sBP) >160 mmHg or diastolic blood pressure (dBP) >100 mmHg measured in the sitting position at Visit 1
* Current active renal disease
* Any history of pyelonephritis
* Evidence of active liver disease
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST) or alkaline phosphatase >2 times the upper limit of the reference range (ULRR), or total bilirubin >1.5 times the ULRR at Visit 1
* Past history of acute pancreatitis with current triglycerides 4.56 mmol/L (400 mg/dL) at Visit 1
* History of malignancy within the past 3 years, other than non-melanoma skin cancer (i.e., basal or superficial squamous cell carcinoma) and treated cervical cancer in-situ
* Any planned major surgery to be performed during the study (e.g., coronary artery bypass surgery, abdominal aortic aneurysm repair, etc.)
* Current life-threatening condition
* Significant hypersensitivity to NSAIDs (e.g., difficulty swallowing or breathing, tachycardia, anaphylaxis, angioedema or skin reaction)
* Pregnancy (defined by positive urine pregnancy test) or lactation at Visit 1, or planning to become pregnant prior to completion of the study
* History or suspicion of alcohol or substance abuse (current or past 6 months).
* Participation in any clinical trial within 30 days prior to Visit 1
* Subjects with a history of hypersensitivity to products containing tiaprofenic acid, suprofen, fenofibrate, oxybenzone, or octocrylene (e.g., sunscreen, perfume)
* Subjects with a history of photosensitivity
* Any clinically significant abnormality or any reason that the subject may not be able to complete the full study observational period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who experience pain relief 2 hours following the first application of ELS-M11 | 2 hours
  Pain relief (as defined by a one point decrease on a 4 point pain intensity scale) in subjects experiencing a moderate to severe migraine headache, 2 hours after the initial application of ELS-M11.

SECONDARY OUTCOMES:
Percentage of patients who report pain relief at various time points within a 24 hour period, following the first application of ELS-M11 | 24 hours
  Pain relief (as defined by a one point decrease on a 0-3 point pain intensity scale) in subjects experiencing a moderate to severe migraine headache over a 24 hour period following the first application of ELS-M11.
Percentage of patients who report complete pain resolution within 24 hours following the first application of ELS-M11. | 24 hours
  Complete resolution (intensity score of 0 on a 0-3 pain scale) of migraine pain within 24 hours, following ELS-M11 application in subjects experiencing a moderate to severe migraine headache.
Percentage of patients who report sustained pain relief after the first application of ELS-M11 | 24 hours
  Sustained pain relief defined as pain relief by 2 hours post study medication application with no increase in the pain intensity score up to 24 hours post medication application in moderate and severe headaches, following ELS-M11 application.
Percentage of patients who report sustained complete pain resolution after the first application of ELS-M11. | 24 hours
  Sustained complete pain resolution defined as pain free by 2 hours post study medication application with no change in a pain intensity score of 0 up to 24 hours post medication application in moderate and severe headaches, following ELS-M11 application.
Time to Initial Use of Rescue Medication following the first application of ELS-M11 | 24 hours
  Time to Initial Use of Rescue Medication following ELS-M11 application in subjects experiencing moderate to severe headaches within a 24 hour period
Use of Rescue Medication following the first application of ELS-M11 by 24 hours | 24 hours
  Use of Rescue Medication within 24 hours following ELS-M11 application in patients experiencing moderate to severe migraine headaches.
Resolution of migraine-associated symptoms, following the first application of ELS-M11 | 24 hours
  Free of migraine-associated symptoms within 24 hours after ELS-M11 application in patients experiencing moderate to severe migraine headaches.
Percentage of patients who can resume or maintain their normal routine, following the first application of ELS-M11. | 24 hours
  Resuming or maintaining normal routine within 24 hours after first study medication application in moderate and severe headaches.

CONTACTS AND LOCATIONS:
Overall Officials: Crist J. Frangakis, Ph.D., Study Chair — Achelios Therapeutics, Inc.
Locations (2):
- United States (2):
  - Michigan Head Pain and Neurological Institute, Ann Arbor, Michigan
  - Coastal Carolina Research Center, Charleston, South Carolina